CLINICAL TRIAL: NCT03422471
Title: Hypoglycemia and Autonomic Nervous System Function
Brief Title: Hypoglycemia and Autonomic Nervous System Function- B2
Acronym: HypoANS-B2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Gail Kurr Adler, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004P001233-B2; R01HL111465 (NIH); K24HL103845 (NIH); UL1TR001102 (NIH); T32HL007609 (NIH)
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Hypoglycemia; Type2 Diabetes
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypoglycemia (Experimental): Participants are exposed to two 90 minute episodes of hypoglycemia (50 mg/dl) through a hyperinsulinemic hypoglycemic clamp. Baroreflex sensitivity will be assessed before, during, and 16 hours after the hypoglycemia.
  Interventions: Other: Hyperinsulinemic Hypoglycemic Clamp

INTERVENTIONS:
Other: Hyperinsulinemic Hypoglycemic Clamp — Participants will receive two 90 minute sessions of hypoglycemia. Baroreflex sensitivity will be assessed before, after, and during the sessions.

SUMMARY:
We will study the effect of hypoglycemia (low blood sugar) on baroreflex sensitivity in participants with well controlled type 2 diabetes.

DETAILED DESCRIPTION:
Participants are admitted for two days and two nights to an inpatient clinical research center for performance of study procedures. On Day 1, two hyperinsulinemic hypoglycemic (50 mg/dl) clamps are performed - an AM clamp from about 9 to 11 am and a PM clamp from about 1 to 3 pm.. Modified Oxford procedures are performed in duplicate at five time points -- before the AM clamp, during the AM clamp, before the PM clamp, during the PM clamp, and the morning of Day 2 (about 16 hrs after completion of the the PM clamp). The Modified Oxford procedure involves the sequential intravenous administration of nitroprusside and phenylephrine with assessment of blood pressure and heart rate by finapress. Baroreflex sensitivity is the relationship of changes in heart rate to changes in blood pressure. .

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18 to 55 years
* Type 2 Diabetes Mellitus controlled by diet, exercise and non-insulin glycemic control agents (metformin, thiazolidinediones, sulfonylureas, dipeptidyl peptidase-4 inhibitors, sodium-glucose co-transporter 2 inhibitors, alpha-glucosidase inhibitors or glucagon-like peptide-1 receptor agonist) or basal insulin at doses less than or equal to 0.3 units/ kg per day.

Exclusion Criteria:

* Hemoglobin A1c > 9% for type 2 diabetes
* Recurrent hypoglycemic episodes within the past month
* BMI < 25 or > 42 (Type 2 diabetes only)
* Pregnancy
* Lactation
* Clinically significant coronary artery, cerebrovascular, or peripheral vascular disease, or presence of systemic illness that might affect autonomic function. Such illnesses include congestive heart failure, renal, pulmonary, hepatic disease, anemia, malignancies, untreated thyroid disease, and alcoholism.
* Current major depressive illness
* In all subjects, any individuals on oral, injected, inhaled or topical corticosteroids within the last year or oral contraceptives within the past 3 months will be excluded.
* Known hypersensitivity to nitroglycerin, nitroprusside and/or phenylephrine.
* Blood pressure > 160/100 mmHg (applies to participants with T2 diabetes)
* Creatinine > 1.5 mg/dL
* Serum potassium >5.2 mmol/L
* Estimated GFR < 50 mL/min
* Use of Viagra, Cialis, and similar drugs within 72 hours of admission.
* Use of beta-blockers or mineralocorticoid receptor antagonists

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Modified Oxford Method Assessment of Baroreflex Function | Time 0 and 16 hours after hyperinsulinemic hypoglycemic clamps
  Change in baroreflex sensitivity between the first assessment (pre-AM clamp on Day 1) and the final assessment (AM of Day 2, about 16 hours after the PM clamp)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Adler, MD/PhD, Principal Investigator — Brigham and Women's Hospital; Roy Freeman, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The data collected will comply with the NIH requirements for timely release and data sharing. Data will be shared in the form of publications and presentations in scientific forums. As the NIH has noted, the investigators reserve the right to keep the data restricted in order to perform the initial analyses for this grant proposal and will continue to use the data for further, but not prolonged, exclusive use. Of note, the sharing of this data will be limited by at least the following issues, some unique to this proposal and some not unique. Some of the data obtained in this study is defined to be sensitive in nature, which may restrict its ability to be shared. Data may only be shared with the approval of our IRB and is limited by HIPPA and any other regulations that may be promulgated during the course of this proposal.
Time Frame: Data will be shared after completion of study and initial publications which we anticipate to be within 18 months of the final participant completing the study protocol.
Access Criteria: Access to this information must be approved by the Partners IRB.

REFERENCES:
- [Derived] Haas AV, Koefoed A, Easly RM, Celli J, Heydarpour M, Bonyhay I, Freeman R, Adler GK. Effect of hypoglycemia on baroreflex sensitivity in individuals with type 2 diabetes: implications for autonomic control of cardiovascular function in diabetes. Clin Auton Res. 2023 Dec;33(6):727-735. doi: 10.1007/s10286-023-00983-5. Epub 2023 Sep 21. PMID 37733159